CLINICAL TRIAL: NCT03178487
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Upadacitinib in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study Evaluating the Safety and Efficacy of Upadacitinib in Adults With Active Ankylosing Spondylitis
Acronym: SELECT-AXIS 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-098; 2017-000431-14 (EudraCT Number)
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Ankylosing Spondylitis (AS)
Keywords: Upadacitinib; ABT-494; Ankylosing Spondylitis (AS); Safety; Efficacy
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upadacitinib 15 mg (Experimental): Participants will receive 15 mg upadacitinib orally once a day for 14 weeks in Period 1 and continue to receive 15 mg upadacitinib orally once a day for an additional 90 weeks in Period 2.
  Interventions: Drug: Upadacitinib
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once a day for 14 weeks in Period 1. In Period 2 participants will receive 15 mg upadacitinib orally once a day for 90 weeks.
  Interventions: Drug: Upadacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Tablet
  Other Names: ABT-494; RINVOQ™
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of upadacitinib in participants with active ankylosing spondylitis (AS) who have had an inadequate response to at least 2 non-steroidal anti-inflammatory drugs (NSAIDs) or intolerance to or a contraindication for NSAIDs, and who are naïve to biologic disease-modifying anti-rheumatic drugs (bDMARD).

DETAILED DESCRIPTION:
This study includes two periods: a 14-week double-blind placebo-controlled period and a 90-week open-label long-term extension period.

Eligible participants were randomly assigned in a 1:1 ratio to receive upadacitinib 15 mg or placebo for 14 weeks in Period 1.

Participants who completed Period 1 received upadacitinib 15 mg for 90 weeks in the extension period.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a clinical diagnosis of ankylosing spondylitis (AS) and meeting the modified New York criteria for AS.
* Participant must have baseline disease activity as defined by having a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4 and a Patient's Assessment of Total Back Pain score >= 4 based on a 0 - 10 numeric rating scale (NRS) at the Screening and Baseline visits.
* Participant has had an inadequate response to at least two nonsteroidal anti-inflammatory drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or participant has an intolerance to or contraindication for NSAIDs as defined by the Investigator.
* If entering the study on concomitant methotrexate (MTX), leflunomide, sulfasalazine (SSZ), and/or hydroxychloroquine, participant must be on a stable dose of MTX (<= 25 mg/week) and/or SSZ (<= 3 g/day) and/or hydroxychloroquine (<= 400 mg/day) or leflunomide (<= 20 mg/day) for at least 28 days prior to the Baseline visit. A combination of up to two background conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) is allowed except the combination of MTX and leflunomide.
* If entering the study on concomitant oral corticosteroids, participant must be on a stable dose of prednisone (<= 10 mg/day), or oral corticosteroid equivalents, for at least 14 days prior to the Baseline visit.
* If entering the study on concomitant NSAIDs, tramadol, combination of acetaminophen and codeine or hydrocodone, and/or non-opioid analgesics, participant must be on stable dose(s) for at least 14 days prior to the Baseline visit.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Prior exposure to any biologic therapy with a potential therapeutic impact on spondyloarthritis (SpA).
* Intra-articular joint injections, spinal/paraspinal injection(s), or parenteral administration of corticosteroids within 28 days prior to the Baseline visit. Inhaled or topical corticosteroids are allowed.
* Participant on any other DMARDs (other than those allowed), thalidomide or apremilast within 28 days or five half-lives (whichever is longer) of the drug prior to the Baseline visit.
* Participant on opioid analgesics (except for combination acetaminophen/codeine or acetaminophen/hydrocodone which are allowed) or use of inhaled marijuana within 14 days prior to the Baseline visit.
* Participant has a history of inflammatory arthritis of different etiology other than axial SpA (including but not limited to rheumatoid arthritis, psoriatic arthritis, mixed connective tissue disease, systemic lupus erythematosus, reactive arthritis, scleroderma, polymyositis, dermatomyositis, fibromyalgia), or any arthritis with onset prior to 17 years of age.
* Laboratory values meeting the following criteria within the Screening period prior to the first dose of study drug: serum aspartate transaminase > 2 × upper limit of normal (ULN); serum alanine transaminase > 2 × ULN; estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease formula < 40 milliliter (mL)/minute/1.73m^2; hemoglobin < 10 gram/deciliter, total white blood cell count < 2,500/microliter (μL); absolute neutrophil count < 1,500/μL; absolute lymphocyte count < 800/μL; and platelet count < 100,000/μL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (101):
- United States (22):
  - Arizona Arthritis & Rheumatolo /ID# 164446, Phoenix, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 165705, Phoenix, Arizona
  - David S. Hallegua MD /ID# 165090, Beverly Hills, California
  - Covina Arthritis Clinic /ID# 165061, Covina, California
  - St. Joseph Health System /ID# 166166, Fullerton, California
  - Global Research Foundation /ID# 165130, Los Angeles, California
  - Rheumatology Center of San Diego /ID# 166167, San Diego, California
  - Colorado Arthritis Associates /ID# 164444, Lakewood, Colorado
  - Bay Area Arthritis and Osteo /ID# 165023, Brandon, Florida
  - LeJenue Research Associates /ID# 165202, Miami, Florida
  - HMD Research LLC /ID# 205172, Orlando, Florida
  - St. Lukes Clinic /ID# 165827, Meridian, Idaho
  - Clinical Investigation Specialists - Skokie /ID# 164385, Skokie, Illinois
  - Henry Ford Health System /ID# 165515, Detroit, Michigan
  - Aa Mrc Llc /Id# 165100, Grand Blanc, Michigan
  - St. Lawrence Health System /ID# 165025, Potsdam, New York
  - DJL Clinical Research, PLLC /ID# 165044, Charlotte, North Carolina
  - Altoona Ctr Clinical Res /ID# 164470, Duncansville, Pennsylvania
  - Clinical Research Ctr Reading /ID# 164876, Wyomissing, Pennsylvania
  - Comprehensive Arthritis Care, a division of Comprehensive Rheumatology Care PLLC /ID# 168107, Hendersonville, Tennessee
  - Diagnostic Group Integrated He /ID# 165195, Beaumont, Texas
  - Arth and Osteo Clin Brazo Valley /ID# 165194, College Station, Texas
- Australia (2):
  - Princess Alexandra Hospital /ID# 169239, Woolloongabba, Queensland
  - Emeritus Research /ID# 169240, Camberwell, Victoria
- Belgium (3):
  - UZ Gent /ID# 166017, Ghent, Oost-Vlaanderen
  - ReumaClinic Genk /ID# 166018, Genk
  - UZ Leuven /ID# 166019, Leuven
- Canada (4):
  - Rheumatology Research Assoc /ID# 165240, Edmonton, Alberta
  - University of Alberta - Division of Rheumatology /ID# 165239, Edmonton, Alberta
  - Credit Valley Rheumatology /ID# 200087, Mississauga, Ontario
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 165238, Sainte-Foy, Quebec
- Croatia (2):
  - Clinical Hospital Dubrava /ID# 167049, Zagreb
  - Medical Center Kuna-Peric /ID# 164851, Zagreb
- Czechia (4):
  - Revmatologicky ustav Praha /ID# 167004, Prague, Praha 2
  - Thomayerova nemocnice /ID# 167003, Prague, Praha 4
  - REVMACLINIC s.r.o. /ID# 167171, Brno
  - ARTHROHELP, s.r.o. /ID# 167001, Pardubice
- Vejle Sygehus /ID# 165190, Vejle, Region Syddanmark, Denmark
- Finland (2):
  - Helsinki Univ Central Hospital /ID# 165794, Helsinki
  - Kiljava Medical Research /ID# 165793, Hyvinkää
- France (3):
  - CHU Bordeaux-Hopital Pellegrin /ID# 166309, Bordeaux
  - CHRU Tours - Hopital Trousseau /ID# 165109, Chambray-lès-Tours
  - CHRU de Montpellier - Hôpital Lapeyronie /ID# 166308, Montpellier
- Germany (4):
  - Rheumazentrum Ruhrgebiet /ID# 165148, Herne, North Rhine-Westphalia
  - Kerckhoff Klinik GmbH /ID# 165158, Bad Nauheim
  - Charite - Campus Benjamin Franklin Medizinische Klinik - Rheumatologie /ID# 165153, Berlin
  - Hamburger Rheuma Forschungszentrum II im MVZ Rheumatologie und Autoimmunmedizin /ID# 165146, Hamburg
- Hungary (4):
  - Revita Reumatologiai Rendelo /ID# 164724, Budapest
  - University of Debrecen /ID# 165674, Debrecen
  - Vita Verum Medical Bt. /ID# 165066, Székesfehérvár
  - Vital Medical Center Orvosi-es Fogaszati Kozpont /ID# 164741, Veszprém
- Italy (4):
  - Ospedale Sant Orsola Malpighi /ID# 165692, Bologna, Emilia-Romagna
  - Policlinico Paolo Giaccone /Id# 165663, Palermo, Sicily
  - ASST G. Pini /ID# 165715, Milan
  - A.O. Universitaria Senese /ID# 165716, Siena
- Japan (17):
  - Hospital of the University of Occupational and Environmental Health /ID# 164380, Kitakyushu-shi, Fukuoka
  - Gunma University Hospital /ID# 165683, Maebashi, Gunma
  - National Hospital Organization Asahikawa Medical Center /ID# 164566, Asahikawa-shi, Hokkaido
  - Kagawa University Hospital /ID# 167517, Kita-gun, Kagawa-ken
  - Kochi Medical School Hospital /ID# 164460, Nankoku-shi, Kochi
  - Shinshu University Hospital /ID# 165304, Matsumoto-shi, Nagano
  - Japanese Red Cross Okayama Hospital /ID# 164376, Okayama, Okayama-ken
  - National Hospital Organization Osaka Minami Medical Center /ID# 164365, Kawachinagano-shi, Osaka
  - Osaka City University Hospital /ID# 165253, Osaka, Osaka
  - Osaka University Hospital /ID# 166033, Suita-shi, Osaka
  - Saitama Medical University Hospital /ID# 164577, Iruma-gun, Saitama
  - Juntendo University Koshigaya Hospital /ID# 165809, Koshigaya-shi, Saitama
  - Tokushima University Hospital /ID# 165108, Tokushima, Tokushima
  - Juntendo University Hospital /ID# 164738, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 165219, Chuo-ku, Tokyo
  - Daido Hospital /ID# 163886, Nagoya
  - Okayama Saiseikai Outpatient Center Hospital /ID# 165595, Okayama
- Netherlands (2):
  - Universitair Medisch Centrum Groningen /ID# 165681, Groningen
  - Medisch Centrum Leeuwarden /ID# 166937, Leeuwarden
- New Zealand (2):
  - Waikato Hospital /ID# 169242, Hamilton, Waikato Region
  - Middlemore Hospital /ID# 169241, Auckland
- Poland (3):
  - Osteo-Medic S.C. /ID# 165646, Bialystok, Podlaskie Voivodeship
  - ETYKA-Osrodek Badan Klinicznyc /ID# 165634, Olsztyn, Warmian-Masurian Voivodeship
  - NZOZ Nasz Lekarz /ID# 166023, Torun
- Portugal (5):
  - Instituto Portugues De Reumatologia /ID# 168314, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 168312, Lisbon, Lisbon District
  - Centro Hospitalar de Vila Nova Gaia/Espinho, EPE /ID# 168313, Vila Nova de Gaia, Porto District
  - Hospital CUF Descobertas /ID# 168311, Lisbon
  - Unidade Local De Saude Do Alto Minho /ID# 168310, Viana do Castelo
- South Korea (7):
  - Chungnam National University Hospital /ID# 164561, Junggu, Daejeon Gwang Yeogsi
  - Gachon University Gil Medical Center /ID# 165114, Incheon, Incheon Gwang Yeogsi
  - Chonnam National University Hospital /ID# 164541, Gwangju, Jeonranamdo
  - Hanyang University Seoul Hospi /ID# 165811, Seongdong-gu, Seoul Teugbyeolsi
  - Cath Univ Seoul St Mary's Hosp /ID# 164549, Seoul, Seoul Teugbyeolsi
  - Kyunghee University Hospital at Gangdong /ID# 164569, Seoul
  - Asan Medical Center /ID# 164557, Seoul
- Spain (3):
  - Hospital Unversitario Marques de Valdecilla /ID# 165028, Santander, Cantabria
  - Hospital Parc de Salut del Mar /ID# 165027, Barcelona
  - Corporac Sanitaria Parc Tauli /ID# 165029, Barcelona
- Sweden (2):
  - Skanes Universitetssjukhus /ID# 165712, Malmo, Skåne County
  - Reumatologkliniken /ID# 165713, Västerås
- United Kingdom (5):
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 166202, Warrington, Cheshire West And Chester
  - Whipps Cross Univ Hospital /ID# 165150, London, London, City of
  - Norfolk and Norwich Univ Hosp /ID# 165149, Norwich, Norfolk
  - Royal National Hosp for Rheuma /ID# 165147, Bath
  - Glasgow Royal Infirmary /ID# 165152, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] van der Heijde D, Song IH, Pangan AL, Deodhar A, van den Bosch F, Maksymowych WP, Kim TH, Kishimoto M, Everding A, Sui Y, Wang X, Chu AD, Sieper J. Efficacy and safety of upadacitinib in patients with active ankylosing spondylitis (SELECT-AXIS 1): a multicentre, randomised, double-blind, placebo-controlled, phase 2/3 trial. Lancet. 2019 Dec 7;394(10214):2108-2117. doi: 10.1016/S0140-6736(19)32534-6. Epub 2019 Nov 12. PMID 31732180
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Navarro-Compan V, Van den Bosch F, Sampaio-Barros PD, Ostor AJK, Parikh B, Kato K, Gao T, Stigler J, Ramiro S. Efficacy of upadacitinib in subgroups of patients with axial spondyloarthritis with early versus established disease. RMD Open. 2025 Mar 4;11(1):e005110. doi: 10.1136/rmdopen-2024-005110. PMID 40037923
- [Derived] Burmester GR, Stigler J, Rubbert-Roth A, Tanaka Y, Azevedo VF, Coombs D, Lagunes I, Lippe R, Wung P, Gensler LS. Safety Profile of Upadacitinib up to 5 Years in Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis: An Integrated Analysis of Clinical Trials. Rheumatol Ther. 2024 Jun;11(3):737-753. doi: 10.1007/s40744-024-00671-4. Epub 2024 Apr 29. PMID 38683479
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Deodhar A, van der Heijde D, Sieper J, Van den Bosch F, Maksymowych WP, Kim TH, Kishimoto M, Ostor A, Combe B, Sui Y, Chu AD, Song IH. Safety and Efficacy of Upadacitinib in Patients With Active Ankylosing Spondylitis and an Inadequate Response to Nonsteroidal Antiinflammatory Drug Therapy: One-Year Results of a Double-Blind, Placebo-Controlled Study and Open-Label Extension. Arthritis Rheumatol. 2022 Jan;74(1):70-80. doi: 10.1002/art.41911. Epub 2021 Nov 12. PMID 34196498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between October 24, 2017, and September 10, 2018 at 62 sites in 20 countries in North America, Eastern and Western Europe, Asia, and Oceania.
  This study consists of a 14-week double-blind treatment period (Period 1) and a 90-week long-term extension period (Period 2) for participants who completed Period 1.
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to one of two treatment groups. Randomization was stratified by screening concentrations of high-sensitivity C-reactive protein (hsCRP; ≤ upper limit of normal [ULN] vs > ULN; where the ULN is 2.87 mg/L) and geographical region (USA and Canada, Japan, rest of the world).
Groups:
- Placebo / Upadacitinib 15 mg: Participants received matching placebo orally once a day for 14 weeks in Period 1. Participants then received upadacitinib 15 mg orally once a day for 90 weeks in Period 2.
- Upadacitinib 15 mg: Participants received 15 mg upadacitinib orally once a day for 14 weeks in Period 1, and continued to receive upadacitinib 15 mg orally once a day for 90 weeks in Period 2.
Period: Period 1
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 15 mg
Started | 94 | 93
Received Treatment | 94 | 93
Completed (Completed Period 1) | 90 | 89
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 0 | 1
Period: Period 2
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 15 mg
Started | 90 | 89
Received Treatment | 89 | 89
Completed | 69 | 70
Not Completed | 21 | 19
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Coronavirus Disease 2019 (COVID-19) Logistical Restrictions | 1 | 0
Not completed — Other | 8 | 7

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) includes all randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received matching placebo orally once a day for 14 weeks in Period 1.
- Upadacitinib 15 mg: Participants received 15 mg upadacitinib orally once a day for 14 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 15 mg | Total
Number analyzed (Participants) | 94 | 93 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.07) | 47.0 (12.78) | 45.4 (12.50)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 39 | 28 | 67
  40 - 64 years | 53 | 56 | 109
  ≥ 65 years | 2 | 9 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 69 | 63 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 89 | 89 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76 | 79 | 155
  Black or African American | 2 | 1 | 3
  Asian | 16 | 13 | 29
Region [Count of Participants; unit: Participants]
  USA and Canada | 10 | 9 | 19
  Western Europe | 33 | 30 | 63
  Eastern Europe | 34 | 36 | 70
  Japan | 7 | 6 | 13
  South Korea | 7 | 6 | 13
  Australia and New Zealand | 3 | 6 | 9
Duration Since Ankylosing Spondylitis (AS) Diagnosis [Mean (Standard Deviation); unit: years] | 6.0 (6.79) | 7.8 (10.64) | 6.9 (8.94)
Duration of Ankylosing Spondylitis Symptoms [Mean (Standard Deviation); unit: years] | 14.0 (9.86) | 14.8 (11.64) | 14.4 (10.76)
Patient's Global Assessment of Disease Activity (PtGA) [Mean (Standard Deviation); unit: units on a scale] — Assessed by the participant using a numeric rating scale (NRS) ranging from 0 (No activity) to 10 (Severe activity). Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 94 | 91 | 185
    (all) | 6.8 (1.66) | 6.6 (1.81) | 6.7 (1.73)
Patient's Assessment of Total Back Pain [Mean (Standard Deviation); unit: units on a scale] — Total back pain was assessed by the participant on a NRS from 0 (no pain) to 10 (most severe pain). Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 94 | 92 | 186
    (all) | 6.7 (1.78) | 6.8 (1.77) | 6.8 (1.78)
Bath Ankylosing Spondylitis Functional Index [Mean (Standard Deviation); unit: units on a scale] — The Bath Ankylosing Spondylitis Functional Index (BASFI) is used to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities, each scored on a NRS ranging from 0 (easy to perform activity) to 10 (impossible to perform activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher score indicating more functional limitations. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 94 | 91 | 185
    (all) | 5.5 (2.17) | 5.4 (2.36) | 5.4 (2.26)
Inflammation [Mean (Standard Deviation); unit: units on a scale] — Inflammation was measured by the mean of the two morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration). Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 94 | 92 | 186
    (all) | 6.7 (1.90) | 6.5 (1.99) | 6.6 (1.94)
High-sensitivity C-reactive Protein (hsCRP) Level at Screening [Count of Participants; unit: Participants] — The Screening level of hsCRP was a randomization stratification factor. The hsCRP upper limit of normal (ULN) = 2.87 mg/L.
  Participants
    > upper limit of normal | 68 | 67 | 135
    ≤ upper limit of normal | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) 40 Response at Week 14
Description: ASAS 40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Week 14
Population: Full analysis set; participants who discontinued study drug prior to Week 14 or with missing data at Week 14 were counted as non-responders (non-responder imputation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 94 | 93
percentage of participants | 25.5 [16.7 to 34.3] | 51.6 [41.5 to 61.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusting for stratification factor of Screening hsCRP level; Response Rate Difference = 26.1, 95% CI 2-sided [12.6 to 39.5] — Response Rate Difference = Upadacitinib - Placebo

2. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 14
Description: ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L.
  The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 14 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 84 | 84
score on a scale | -0.54 [-0.71 to -0.37] | -1.45 [-1.62 to -1.28]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeated Measurement; MMRM model includes treatment, visit, treatment-by-visit interaction as fixed effects and Screening hsCRP level and Baseline value as covariates; Least Squares (LS) Mean Difference = -0.91, 95% CI 2-sided [-1.14 to -0.68] — Treatment difference = Upadacitinib - Placebo

3. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Score for the Spine at Week 14
Description: In the SPARCC MRI assessment of the spine, the entire spine is evaluated for active inflammation (bone marrow edema). Six discovertebral units (DVU) representing the 6 most abnormal DVUs were selected to calculate the MRI Spine SPARCC score. For each of the 6 DVUs, 3 consecutive sagittal slices were assessed in 4 quadrants to evaluate the extent of inflammation in all three dimensions.
  Each quadrant was scored for the presence (1) or absence (0) of edema. If edema was present in at least one quadrant of a DVU slice, it was also scored for intensity and depth of the edema representing that slice: An additional score of 1 was assigned if an intense signal was seen in any quadrant on a DVU slice. Slices that included a lesion demonstrating continuous increased signal of depth ≥ 1 cm extending from the endplate were scored as an additional 1 per slice.
  The maximum (worst) overall score for all 6 DVUs is 108.
Time Frame: Baseline and Week 14
Population: Full analysis set; the following MRI data were included in the analysis: Baseline includes MRI data up to 3 days post first dose of study drug and Week 14 includes MRI data up to first dose of period 2 study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 60 | 68
score on a scale | -0.22 [-2.01 to 1.57] | -6.93 [-8.58 to -5.28]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA; ANCOVA model including treatment and Screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -6.71, 95% CI 2-sided [-9.01 to -4.41] — Treatment difference = Upadacitinib - Placebo

4. Secondary Outcome: Percentage of Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response at Week 14
Description: The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For Questions 1 to 5 (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from Baseline in BASDAI score.
Time Frame: Baseline and Week 14
Population: Full analysis set; non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 94 | 93
percentage of participants | 23.4 [14.8 to 32.0] | 45.2 [35.0 to 55.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including BASDAI 50; within the group, the allocated α was adjusted based on the magnitude of p values; p = 0.002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for stratification factor of Screening hsCRP level; Response Rate Difference = 21.8, 95% CI 2-sided [8.5 to 35.0] — Response rate difference = Upadacitinib - Placebo

5. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score
Description: The ASQoL consists of 18 items related to quality of life, including the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. Each item is answered as yes (scored as 1) or no (scored as 0).
  Scores are summed to obtain the overall score which ranges from 0 to 18, where higher scores indicate a worse quality of life. A negative change from Baseline in ASQoL indicates improvement in quality of life.
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 88 | 88
score on a scale | -2.67 [-3.58 to -1.75] | -4.20 [-5.12 to -3.29]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including ASQoL; within the group, the allocated α was adjusted based on the magnitude of p values; p = 0.016, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.54, 95% CI 2-sided [-2.78 to -0.30] — Treatment difference = Upadacitinib - Placebo

6. Secondary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) Partial Remission
Description: ASAS partial remission (PR) is defined as an absolute score of ≤ 2 units on a 0 to 10 scale for each of the four following domains:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Week 14
Population: Full analysis set; non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 94 | 93
percentage of participants | 1.1 [0.0 to 3.1] | 19.4 [11.3 to 27.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including ASAS PR; within the group, the allocated α was adjusted based on the magnitude of p values; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for stratification factor of Screening hsCRP level; Response Rate Difference = 18.3, 95% CI 2-sided [10.0 to 26.6] — Response rate difference = Upadacitinib - Placebo

7. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 14
Description: The Bath Ankylosing Spondylitis Functional Index is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities such as putting on socks, bending, reaching, getting up from the floor or an armless chair, standing, climbing and other physical activities. Each item is scored on a NRS ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. A negative change from Baseline in BASFI indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 86 | 86
score on a scale | -1.30 [-1.74 to -0.86] | -2.29 [-2.73 to -1.85]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including BASFI; within the group, the allocated α was adjusted based on the magnitude of p values; p = 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.00, 95% CI 2-sided [-1.60 to -0.39] — Treatment difference = Upadacitinib - Placebo

8. Secondary Outcome: Change From Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMI[Lin]) at Week 14
Description: The BASMI is a composite score based on 5 direct measurements of spinal mobility:
  1. cervical rotation (measured in degrees),
  2. tragus to wall distance (in centimeters [cm])
  3. lumbar side flexion (in cm),
  4. lumbar flexion (modified Schober's) (in cm) and
  5. intermalleolar distance (in cm).
  Each measurement is converted to a linear score between 0 and 10. The total BASMI score is the average of the 5 scores and ranges from 0 to 10; the higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 89 | 89
score on a scale | -0.14 [-0.29 to 0.01] | -0.37 [-0.52 to -0.21]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including BASMI(lin); within the group, the allocated α was adjusted based on the magnitude of p values; p = 0.030, ANCOVA; ANCOVA model including treatment and Screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -0.22, 95% CI 2-sided [-0.43 to -0.02] — Treatment difference = Upadacitinib - Placebo

9. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 14
Description: The MASES evaluation was conducted to assess the presence or absence of enthesitis (inflammation of the entheses, or sites where tendons or ligaments insert into the bone) at 13 different sites (first costochondral joint left/right, seventh costochondral joint left/right, posterior superior iliac spine left/right, anterior superior iliac spine left/right, iliac crest left/right, fifth lumbar spinous process, and proximal insertion of Achilles tendon left/right. Each site was scored for presence (1) or absence (0) of enthesitis. The MASES is the sum of the 13 site scores, and ranges from 0 to 13, with higher scores indicating more inflammation of the entheses.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with Baseline enthesitis; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 14 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 51 | 50
score on a scale | -1.41 [-2.02 to -0.80] | -2.25 [-2.86 to -1.64]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including MASES; within the group, the allocated α was adjusted based on the magnitude of p values; p = 0.049, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.84, 95% CI 2-sided [-1.68 to -0.00] — Treatment difference = Upadacitinib - Placebo

10. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Overall Work Impairment at Week 14
Description: The Work Productivity and Activity Impairment Questionnaire: Axial Spondyloarthritis, Version 2.0 (WPAI-Axial Spondyloarthritis) measures the effect of overall health and specific symptoms on productivity at work and outside of work. It consists of 6 questions. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity. Overall Work Impairment indicates the percentage of overall work impairment due to health problems. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis participants who were employed and with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: percent impairment
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 53 | 55
percent impairment | -12.60 [-19.04 to -6.15] | -18.11 [-24.73 to -11.50]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. The testing sequence included a group of endpoints tested by the Hochberg procedure, including WPAI; within the group, the allocated α was adjusted based on the magnitude of p values; p = 0.190, ANCOVA; ANCOVA model including treatment and Screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -5.52, 95% CI 2-sided [-13.82 to 2.78] — Treatment difference = Upadacitinib - Placebo

11. Secondary Outcome: Change From Baseline in ASAS Health Index (HI) at Week 14
Description: The ASAS HI measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. Each of the 17 questions is answered by the participant as "I agree" (score = 1) or "I disagree" (score = 0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, where a higher score indicates a worse health status. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 88 | 88
score on a scale | -1.38 [-2.11 to -0.65] | -2.75 [-3.48 to -2.02]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other — To preserve the overall type I error rate at α=0.05 level, a step-down approach was used to test the primary and multiplicity-controlled key secondary endpoints. The testing began with the primary endpoint at α=0.05 and continued conditional on significance of higher-ranked endpoint. ASAS HI was to be evaluated only if the group of endpoints tested by Hochberg procedure were all significant; p = 0.007, Mixed Effect Model Repeated Measurement — This comparison was not tested for statistical significance because the hierarchical testing procedures stopped during the Hochberg procedure; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.37, 95% CI 2-sided [-2.37 to -0.37] — Treatment difference = Upadacitinib - Placebo

12. Secondary Outcome: Percentage of Participants Achieving an ASAS 20 Response at Week 14
Description: ASAS 20 response was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 1 unit (on a scale of 0 to 10) from Baseline in at least 3 of the following 4 domains, with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 units [on a scale of 0 to 10]) in the remaining domain:
  * Patient's global assessment of disease activity, measured on a NRS from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the BASFI which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related BASDAI NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Week 14
Population: Full analysis set; non-responder imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 94 | 93
percentage of participants | 40.4 [30.5 to 50.3] | 64.5 [54.8 to 74.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p = 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusting for stratification factor of Screening hsCRP level; Response Rate Difference = 24.1, 95% CI 2-sided [10.2 to 38.0]; Response Rate Difference = Upadacitinib - Placebo

13. Secondary Outcome: Change From Baseline in SPARCC MRI Score for Sacroiliac Joints at Week 14
Description: In the SPARCC MRI assessment of the sacroiliac (SI) joints 6 consecutive sacroiliac joint image coronal slices representing the largest proportion of the synovial compartment of the SI joints were assessed for edema, intensity and depth of edema.
  Each SI joint (left and right) was divided into quadrants for a total of 8 SI scoring locations. Each quadrant was scored for the presence (1) or absence (0) of edema, intensity of edema (a score of 1 was assigned for each SI joint (left and right) if an intense signal was seen in any quadrant of that joint for each slice), and a lesion was graded as deep (score of 1) if there was homogeneous and unequivocal increase in signal extending over a depth of at least 1 cm from the articular surface of the SI joint in any quadrant.
  The total maximum score for all SI joints across 6 slices is 72.
Time Frame: Baseline and Week 14
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 59 | 68
score on a scale | -0.22 [-1.47 to 1.04] | -3.91 [-5.05 to -2.77]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p < 0.001, ANCOVA — This comparison was not part of the pre-specified multiplicity testing sequence; ANCOVA model including treatment and Screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -3.69, 95% CI 2-sided [-5.31 to -2.08] — Treatment difference = Upadacitinib - Placebo

14. Post Hoc Outcome: Change From Baseline in SPARCC MRI Score for the Spine at Week 14 - Supplementary Analysis
Description: In the SPARCC MRI assessment of the spine, the entire spine is evaluated for active inflammation (bone marrow edema). Six DVUs representing the 6 most abnormal DVUs were selected to calculate the SPARCC MRI spine score. For each DVU, 3 consecutive sagittal slices were assessed in 4 quadrants to evaluate the extent of inflammation in all dimensions. Each quadrant was scored for the presence (1) or absence (0) of edema. If edema was present in at least 1 quadrant of a DVU slice, it was also scored for intensity and depth of the edema representing that slice: An additional score of 1 was assigned if an intense signal was seen in any quadrant on a DVU slice. Slices that included a lesion demonstrating continuous increased signal of depth ≥ 1 cm extending from the endplate were scored as an additional 1 per slice. The maximum (worst) overall score for all 6 DVUs is 108.
  A supplemental post-hoc SPARCC MRI analysis included all MRI data collected at nominal visits at Baseline and Week 14.
Time Frame: Baseline and Week 14
Population: Full analysis set; the analysis includes all participants with available MRI data collected at Baseline and Week 14
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 88 | 89
score on a scale | -0.65 [-2.20 to 0.90] | -6.86 [-8.41 to -5.30]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p < 0.001, ANCOVA; ANCOVA model including treatment and Screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -6.21, 95% CI 2-sided [-8.27 to -4.14] — Treatment difference = Upadacitinib - Placebo

15. Post Hoc Outcome: Change From Baseline in SPARCC MRI Score for Sacroiliac Joints at Week 14 - Supplementary Analysis
Description: In the SPARCC MRI assessment of the sacroiliac joints 6 consecutive sacroiliac joint image coronal slices representing the largest proportion of the synovial compartment of the SI joints were assessed for edema, intensity and depth of edema.
  Each SI joint (left and right) was divided into quadrants for a total of 8 SI scoring locations. Each quadrant was scored for the presence (1) or absence (0) of edema, intensity of edema (a score of 1 was assigned for each SI joint (left and right) if an intense signal was seen in any quadrant of that joint for each slice), and a lesion was graded as deep (score of 1) if there was homogeneous and unequivocal increase in signal extending over a depth of at least 1 cm from the articular surface of the SI joint in any quadrant. The total maximum score for all SI joints across 6 slices is 72.
  A supplemental post-hoc SPARCC MRI analysis was done to include all MRI data collected at nominal visits at Baseline and Week 14.
Time Frame: Baseline and Week 14
Population: Full analysis set; the analysis includes all participants with available MRI data collected at Baseline and Week 14
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 87 | 89
score on a scale | -0.90 [-2.01 to 0.20] | -3.45 [-4.54 to -2.36]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Other; p < 0.001, ANCOVA; ANCOVA model including treatment and Screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -2.55, 95% CI 2-sided [-4.01 to -1.08] — Treatment difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: Period 1: From the first dose of study drug up to Week 14 or up to 30 days after last dose for participants who discontinued study drug prior to Week 14. Period 1+2: From Week 14 to 30 days after last dose (up to 94 weeks) for participants initially assigned to placebo; From Week 1 up to 30 days after last dose (up to 108 weeks) for participants initially assigned to upadacitinib.
Groups:
- Period 1: Placebo: Participants received matching placebo orally once a day for 14 weeks in Period 1.
- Period 1: Upadacitinib 15 mg: Participants received 15 mg upadacitinib orally once a day for 14 weeks in Period 1.
- Period 1 + 2: Upadacitinib 15 mg: Participants originally assigned to placebo received upadacitinib 15 mg from Week 14 to Week 104. Participants originally assigned to upadacitinib received upadacitinib 15 mg from Week 0 to Week 104.
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 15 mg | Period 1 + 2: Upadacitinib 15 mg
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/93 | 0/182
Serious Adverse Events (participants affected / at risk) | 1/94 | 1/93 | 16/182
Other Adverse Events (participants affected / at risk) | 21/94 | 26/93 | 104/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=94) | Period 1: Upadacitinib 15 mg (N=93) | Period 1 + 2: Upadacitinib 15 mg (N=182)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS NONINFECTIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HEMIPARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
AORTIC DILATATION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=94) | Period 1: Upadacitinib 15 mg (N=93) | Period 1 + 2: Upadacitinib 15 mg (N=182)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 5 (5) | 13 (14)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 1 (1) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 5 (6) | 35 (48)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 23 (30)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 5 (5) | 13 (14)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 8 (8) | 29 (35)
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 13 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 11 (11)
HEADACHE (Nervous system disorders) | 2 (2) | 5 (5) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03178487/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03178487/SAP_001.pdf